CLINICAL TRIAL: NCT03338504
Title: Determining the Mechanism of Myocardial Injury and Role of Coronary Disease in Type 2 Myocardial Infarction
Acronym: DEMAND-MI
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: British Heart Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: FS/16/75/32533
Record Dates: First submitted 2017-11-07; First posted 2017-11-09 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Myocardial Infarction, Acute; Myocardial Ischemia; Myocardial Injury
Keywords: type 2 myocardial infarction
MeSH Terms: conditions — Myocardial Infarction; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma samples will be stored at multiple time points during admission.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Suspected type 2 myocardial infarction: The investigators will identify consecutive patients with acute myocardial injury (defined as a rise and or fall in cardiac troponin concentration on serial testing, with at least one value >99th centile) where the likely mechanism of injury is thought to be myocardial oxygen supply and demand imbalance (e.g secondary to hypoxia, hypotension, tachycardia or anaemia). Patients will be identified through screening of cardiac troponin measurements. Patients who meet both the inclusion and exclusion criteria, will be approached and those who provide consent will comprise the study population. All patients will have a Cardiac MRI scan, with invasive coronary angiography or CT coronary angiography dependent on baseline fitness. The investigators will record demographic and clinical information from the electronic patient record for patients who meet inclusion criteria but have one or more exclusion criteria.
  Interventions: Diagnostic Test: Invasive coronary angiography; Radiation: CT coronary angiography; Diagnostic Test: Cardiac MRI

INTERVENTIONS:
Diagnostic Test: Invasive coronary angiography — Where patients are fit, coronary angiography will be performed via the femoral or radial artery with 6F arterial catheters. In patients with one or more stenoses in a major epicardial vessel, a coronary pressure guidewire (PressureWire™ Aeris™, St. Jude Medical, St. Paul, Minnesota) will be used to determine distal coronary pressure and the fractional flow reserve (FFR) calculated at maximal adenosine-induced (intravenous 140 μg/kg/min) hyperaemia. Optical coherence tomography (OCT) will be performed in all three coronary vessels using a Dragonfly® coronary imaging catheter (Abbott Diagnostics, Abbott Park, Illinois) with pullback at 20 mm/s to identify features consistent with vulnerable plaque or recent plaque rupture.(16) If there is evidence of inducible myocardial ischaemia due to coronary artery stenosis, revascularisation with percutaneous coronary intervention may be considered if in the patients best interests.
Radiation: CT coronary angiography — CT coronary angiography will be performed using a 128 multidetector row CT. Patients with a heart rate exceeding 65 beats/min will receive oral beta-blockade 1 hour before computed tomography. Additional intravenous beta blockers will be given depending on heart rate at the time of imaging. All patients will receive sublingual glyceryl trinitrate (300 μg) immediately prior to dual cardiac and respiratory-gated computed tomography imaging of the coronary arteries. The investigators will quantify total plaque burden using CT calcium scoring. A bolus of 80-100 mL of contrast will be injected intravenously at 5 mL/s. An assessment of the functional consequences of coronary artery stenosis will be made using the computed tomography fractional flow reserve (CT-FFR) technique, using the HeartFlow platform.
Diagnostic Test: Cardiac MRI — Cardiovascular magnetic resonance (CMR) will be performed using a 3T scanner. The MRI scan will consist of localisers, axial and coronal HASTE images, standard breath-held and ECG-gated cine sequences. Short-axis cine images will be obtained for the assessment of left ventricle function and volumes. Left ventricle volumes, mass and ejection fraction will be assessed using dedicated software and values indexed to body surface area. Breath-held, ECG-gated T2 mapping sequences of the myocardium will be performed in the short-axis as a marker of myocardial inflammation. T1-weighted imaging of the coronary arteries will be performed to look for evidence of recent intraplaque thrombus or haemorrhage. The late gadolinium enhancement and T2 mapping techniques will identify regions of new or old myocardial infarction as well as other patterns of injury. Where there are no contraindications, stress MRI will be performed using intravenous Regadenoson.

SUMMARY:
Myocardial injury is common in patients without acute coronary syndrome, and therefore international guidelines propose a classification of patients with myocardial infarction by aetiology. This differentiates between myocardial infarction due to plaque rupture (type 1) and myocardial oxygen supply-demand imbalance (type 2) in other acute illnesses. However, these guidelines have not been widely adopted as the diagnostic criteria for type 2 myocardial infarction are not clearly defined. Patients with type 2 myocardial infarction have poor long term outcomes, with at least twice the mortality at five years compared to those with an index type 1 myocardial infarction. Despite the majority of deaths being attributable to non-cardiovascular events, the rate of future type 1 myocardial infarction or cardiovascular death is similar regardless of index classification. If this future risk is related to the presence of underlying coronary artery disease, then there may be the potential to improve outcomes through targeted investigation and secondary prevention. The investigators will undertake a systematic evaluation of the mechanism of myocardial injury and the role of coronary artery disease in 100 patients with elevated cardiac troponin concentrations where the diagnosis is likely to be type 2 myocardial infarction. These studies will help improve the assessment of patients with myocardial injury, refine the diagnostic criteria for type 2 myocardial infarction, and aid the design of future therapeutic trials.

DETAILED DESCRIPTION:
The investigators will systematically evaluate the mechanisms of acute myocardial injury in unselected patients who present to hospital with an alternative primary illness likely to cause myocardial oxygen supply or demand imbalance. All patients will be assessed by a member of the study team during their index admission and will undergo a detailed assessment of their coronary anatomy with either computed tomography coronary angiography (CTCA), CT calcium scoring and non-invasive fractional flow reserve assessment (CT-FFR) or invasive coronary angiography with optical coherence tomography (OCT) and invasive fractional flow reserve (FFR). The pattern of myocardial injury and its functional consequence will be evaluated by cardiac magnetic resonance (CMR) imaging. The investigators will determine the kinetics of cardiac troponin release using serial testing at multiple time points throughout admission, and quantify other proteins and the expression of long non-coding RNA and associated mRNA to identify differences related to the presence of coronary artery disease, which may help to identify new biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Unscheduled hospital admission with acute myocardial injury (defined as a rise and or fall in high-sensitivity cardiac troponin I concentrations on blood testing)
* A suspected aetiology of myocardial oxygen supply and demand imbalance with symptoms or signs of myocardial ischaemia

Exclusion Criteria:

* Unable or unwilling to give informed consent
* Women who are pregnant, breastfeeding or of child-bearing potential (women who have experienced menarche, are pre-menopausal and have not been sterilised) will not be enrolled into the trial.
* Probable type 1 myocardial infarction
* Renal impairment (estimated glomerular filtration rate ≤30ml/min/1.73m2)
* Severe hepatic impairment
* Frailty with inability to self-transfer (determined using Katz Index)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospitalized patients with acute myocardial injury (defined as a rise and or fall in cardiac troponin concentration on serial testing, with at least one value >99th centile) where the likely mechanism of injury is thought to be myocardial oxygen supply and demand imbalance (e.g secondary to hypoxia, hypotension, tachycardia or anaemia).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2021-11-06 (Actual)

PRIMARY OUTCOMES:
Prevalence of coronary disease | 30 days of index presentation
  Defined as obstructive (if stenosis >50% in the left main stem or >70% in a major epicardial vessel) or non obstructive disease

SECONDARY OUTCOMES:
Lesion severity | 30 days of index presentation
  Assessed using the invasive (FFR) or non-invasive (CT-FFR) fractional flow reserve technique
Presence of intraluminal plaque rupture | 30 days of index presentation
  Determined using invasive optical coherence tomography
Pattern of myocardial injury | 30 days of index presentation
  Determined using the late gadolinium enhancement technique
Cardiovascular death and future myocardial infarction | 1 year
  We will determine prevalence of major adverse cardiovascular events at one year in the study population, and those screened but not eligible for recruitment, to ensure a representative cohort.
All cause mortality | 1 year
  We will determine prevalence of major adverse cardiovascular events at one year in the study population, and those screened but not eligible for recruitment, to ensure a representative cohort.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Cardiovascular Science, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Requests for IPD will be considered on an individual basis.

REFERENCES:
- [Background] Chapman AR, Adamson PD, Mills NL. Assessment and classification of patients with myocardial injury and infarction in clinical practice. Heart. 2017 Jan 1;103(1):10-18. doi: 10.1136/heartjnl-2016-309530. Epub 2016 Nov 2. PMID 27806987
- [Derived] Boeddinghaus J, Bularga A, Taggart C, Wereski R, McDermott M, Thurston AJF, Ferry AV, Williams MC, Baker AH, Dweck MR, Newby DE, Chapman AR, Lindahl B, Mills NL; DEMAND-MI Investigators. Implications of a new clinical classification of acute myocardial infarction. Eur Heart J Acute Cardiovasc Care. 2025 Mar 22;14(3):131-141. doi: 10.1093/ehjacc/zuaf002. PMID 39824208
- [Derived] Meah MN, Bularga A, Tzolos E, Chapman AR, Daghem M, Hung JD, Chiong J, Taggart C, Wereski R, Gray A, Dweck MR, Roobottom C, Curzen N, Kardos A, Felmeden D, Mills NL, Slomka PJ, Newby DE, Dey D, Williams MC. Distinguishing Type 1 from Type 2 Myocardial Infarction by Using CT Coronary Angiography. Radiol Cardiothorac Imaging. 2022 Oct 27;4(5):e220081. doi: 10.1148/ryct.220081. eCollection 2022 Oct. PMID 36339063
- [Derived] Bularga A, Hung J, Daghem M, Stewart S, Taggart C, Wereski R, Singh T, Meah MN, Fujisawa T, Ferry AV, Chiong J, Jenkins WS, Strachan FE, Semple S, van Beek EJR, Williams M, Dey D, Tuck C, Baker AH, Newby DE, Dweck MR, Mills NL, Chapman AR. Coronary Artery and Cardiac Disease in Patients With Type 2 Myocardial Infarction: A Prospective Cohort Study. Circulation. 2022 Apr 19;145(16):1188-1200. doi: 10.1161/CIRCULATIONAHA.121.058542. Epub 2022 Mar 28. PMID 35341327